CLINICAL TRIAL: NCT05069376
Title: Effect of Ureteral Stents Length and Location on Related Symptom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Chen-Hsun Ho, Doctor, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N201802031
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Lower Urinary Tract Symptoms; Overactive Bladder Syndrome
Keywords: Ureteral stent; OAB
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Arm 1: Intra-ureteral placement of double-J stent Arm 2: Conventional placement of double-J stent
Who Masked: Participant
Masking Description: Patients were not informed the allocation until the stent was removed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- The intraureteral placement of distal end of ureteral stent (Experimental): Patients randomized to this group received 5-16/5-18 D-J stent with intraureteral placement of the distal end
  Interventions: Device: Ureteral Stent of 5-16 or 5-18
- The conventional placement of the distal end of ureteral stent (Active Comparator): Patients randomized to this group received 5-22/5-24 D-J stent with bladder placement of the distal end
  Interventions: Device: Ureteral Stent of 5-22 or 5-24

INTERVENTIONS:
Device: Ureteral Stent of 5-16 or 5-18 — Boston Scientific Polaris™ Ultra Ureteral Stent
  Arms: The intraureteral placement of distal end of ureteral stent
Device: Ureteral Stent of 5-22 or 5-24 — Boston Scientific Polaris™ Ultra Ureteral Stent
  Arms: The conventional placement of the distal end of ureteral stent

SUMMARY:
This is a prospective randomized clinical trial, evaluating the effect of the intra-ureteral placement of the stent's distal end versus the conventional stent placement on the postoperative LUTS and pain.

DETAILED DESCRIPTION:
Intravesical stent mass has been considered to cause stent-related symptoms, such as LUTS and pain. The current study hypothesized that the total intra-ureteral placement of the stent's distal end could decrease postoperative LUTS and pain. We proposed a prospective randomized trials, investigating the effect of intra-ureteral stent placement versus conventional stent placement. The primary end point was postoperative LUTS. The secondary end points were postoperative pain and quality of life. We used USSQ questionnaire as the assessing tool.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of unilateral ureteral stone
* Plan to undergo unilateral URS lithotripsy
* Adult patients (>18 years old)

Exclusion Criteria:

* Pre-stented cases
* Distal ureteral stones
* Preoperative urinary tract infection
* With medications known to influence stent-related symptoms, including alpha-blockers, antimuscarinics, beta3-agonist
* Pregnancy
* Other procedures required during the procedure of lithotripsy
* A stent was expected to be indwelled for more than 10 days (ureteral stricture, ureteral tumors/polyps, ureteral trauma, and a large amount of stone fragments)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Lower urinary tract symptom after placement of D-J stent | Before removal of D-J stent
  The symptoms are evaluated by a complete USSQ (Ureteral Stent Symptom Questionnaire) urinary index. The minimum and maximum values are 11 and 53, and the higher scores mean a worse outcome

SECONDARY OUTCOMES:
Pain after placement of D-J stent | Before removal of D-J stent
  The symptoms are evaluated by a complete USSQ (Ureteral Stent Symptom Questionnaire) pain index and general health index. The minimum and maximum values of the body pain index are 2 and 43. The minimum and maximum values of the general health index are 4 and 28. The higher scores of both mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hsun Ho, MD, PhD, Principal Investigator — Shuang Ho Hospital Taipei Medical University
Locations (1):
- Shuang Ho Hospital Taipei Medical University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No